CLINICAL TRIAL: NCT00471991
Title: Monocenter, Open-label, Randomized Study to Determine the Ovulation Inhibitory Effect of the Combined Oral Contraceptive SH T04769G and SH D00659AF (0.03 mg Ethinylestradiol and 2.0 mg Dienogest), Applied for Two Treatment Cycles to 60 Healthy Female Volunteers
Brief Title: Valette (Combined Oral Contraceptive SH T04769G and SH D00659AF) Low Ovulation Inhibition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare AG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91539; 2006-006633-41 (EudraCT Number); 310723 (Other: company internal)
Record Dates: First submitted 2007-05-09; First posted 2007-05-10 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Oral Contraceptive
Keywords: Oral contraceptive; ovulation inhibitory effect
MeSH Terms: interventions — Ethinyl Estradiol; dienogest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: SH T04769G
- Arm 2 (Experimental)
  Interventions: Drug: Ethinyl estradiol / dienogest (SH D00659 AF)

INTERVENTIONS:
Drug: SH T04769G — The study consists of 4 cycles resulting in approx. 16 weeks of study participation. The investigational product is an oral contraceptive. 21 tablets are taken each cycle followed by a 7-day tablet-free interval. (One cycle lasts for 28 days.)Volunteers will have to come for a visit every 2 to 4 days over the whole study period.The function of the ovaries is studied by transvaginal ultrasonography and determination of hormonal parameters from blood samples. The mouth of the uterus is inspected during each visit and the cervical smear will be investigated. Adverse events will be recorded and diary entries will be controlled by the investigator.
  Arms: Arm 1
Drug: Ethinyl estradiol / dienogest (SH D00659 AF) — The study consists of 4 cycles resulting in approx. 16 weeks of study participation. The investigational product is an oral contraceptive. 21 tablets are taken each cycle followed by a 7-day tablet-free interval. (One cycle lasts for 28 days.)Volunteers will have to come for a visit every 2 to 4 days over the whole study period.The function of the ovaries is studied by transvaginal ultrasonography and determination of hormonal parameters from blood samples. The mouth of the uterus is inspected during each visit and the cervical smear will be investigated. Adverse events will be recorded and diary entries will be controlled by the investigator.Volunteers have to undergo a series of blood sampling during the 2nd treatment cycle to evaluate the pharmacokinetic (liberation, absorption, distribution, metabolization and excretion) of the new oral contraceptive.
  Arms: Arm 2

SUMMARY:
The aim of this monocenter, open-label, randomized study is to determine the ovulation inhibitory effect of the combined oral contraceptive (COC) SH T04769G and to collect supplementary data regarding the ovulation inhibitory effect of the COC Valette® SH D00659AF (0.03 mg EE and 2.0 mg DNG), each applied for two treatment cycles in 60 healthy female volunteers, aged 18-35 years.Combined oral contraceptives consist of two components: an estrogen and a progestin. The estrogen is required for a regular cycle; the progestin ensures the protection against unwanted pregnancy. In a sufficient dosage, progestins prevent ovulation. The investigational product is an oral contraceptive that contains the estrogen ethinylestradiol and the progestin dienogest as active ingredients. 21 tablets are taken each cycle followed by a 7-day tablet-free interval. Thus, the whole cycle lasts for 28 days.The marketed oral contraceptive Valette® contains both ingredients (ethinylestradiol and dienogest) in a higher dose. One half of the volunteers (30 volunteers) will receive this product. Efficacy and safety were already confirmed by numerous clinical studies.Another 30 volunteers will receive the investigational product. The dose reduction is not assumed to have a negative impact on tolerance.The study is aimed to show whether the reduced dosage is sufficient for contraception.Course of the study:The study consists of 4 cycles (one cycle before treatment, followed by two treatment cycles and one post-treatment cycle) resulting in approx. 16 weeks of study participation. The post-treatment cycle is aimed to observe the return to the normal function of the ovaries. Volunteers will have to come for a visit every 2 to 4 days over the whole study period.Visit 1The investigator will explain the study in detail and the volunteer will be given ample time and opportunity to ask questions. If all questions were answered the volunteer will decide on participation in the study. If she decides to take part, she will give her written consent on the Informed Consent Form.Afterwards, a pregnancy test will be performed, a complete medical, surgical and medication history will be recorded and physical and gynaecological examinations will be performed. Transvaginal ultrasonography will be done and smear from the mouth of the uterus is taken for precaution of cancer.Blood (10 ml) will be drawn to determine routine safety lab, heart rate and blood pressure will be measured and height and weight will be recorded.Volunteers will be provided with a diary that has to be filled in on a daily basis during the whole study period (bleeding records, intake of study medication, performance of pregnancy tests).During the whole study non-hormonal methods of contraception have to be used (condom plus spermicide; diaphragm with spermicide). During the cycle before study treatment, the function of the ovaries is studied by transvaginal ultrasonography and determination of hormonal parameters from blood samples. The mouth of the uterus is inspected during each visit and the cervical smear will be investigated. Visits will be performed every 4 days.If ovulation can be confirmed, volunteers will be randomized to one of the treatment groups.Volunteers who will receive the investigational product will undergo a blood sampling on a given day of this cycle to determine the baseline hormonal status (fasting condition).A home pregnancy test has to be done by the volunteer before intake of the study medication. Only in case a pregnancy is excluded, intake of study medication will start.Treatment cycles:During these cycles, visits are performed every 3 days to determine ovarian activity (transvaginal ultrasonography, blood sampling, inspection of the mouth of the uterus and cervical smear investigation). Adverse events will be recorded and diary entries will be controlled by the investigator.Volunteers who receive the investigational product have to undergo a series of blood sampling during the 2nd treatment cycle to evaluate the pharmacokinetic (liberation, absorption, distribution, metabolization and excretion) of the new oral contraceptive.Post-treatment cycle:Non-hormonal contraceptive methods have also to be used during the post-treatment cycle. It starts immediately after the 2nd treatment cycle, i.e., on the 8th day after the last tablet intake and ends with the start of the next menstrual bleeding. Visits will be performed every 4 days to determine the return of ovarian activity by transvaginal ultrasound measures and blood sampling for hormone determination. After end of the next menstrual bleeding, a final Visit including physical and gynaecological examinations will be performed. Options for further contraceptive methods will be discussed with the investigator.

DETAILED DESCRIPTION:
The trial is sponsored by Bayer Schering Pharma AG, Germany.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers, aged 18 - 35 years (smokers up to 30 years)
* Willingness to apply non-hormonal methods of contraception during the course of the study (e.g., condom with spermicide, diaphragm with spermicide)
* Confirmation of ovulation during the cycle before treatment
* Normal routine blood values

Exclusion Criteria:

* Contraindications for the use of oral contraceptives
* Pregnancy, lactation
* Simultaneous participation in another clinical study
* Considerable overweight

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable is ovulation inhibition in Cycle 2 (yes/no). Ovarian activity will be classified according to Hoogland and Skouby (1993). | 4 cycles: one cycle before treatment followed by two treatment cycles (28 days each, 21 days with tablet intake followed by a 7-day tablet-free interval) one post-treatment cycle

SECONDARY OUTCOMES:
Follicle size (leading follicle) by transvaginal ultrasonography | 4 cycles: one cycle before treatment followed by two treatment cycles (28 days each, 21 days with tablet intake followed by a 7-day tablet-free interval) one post-treatment cycle
Endogenous hormones (estradiol, progesterone, FSH, LH) | 4 cycles: one cycle before treatment followed by two treatment cycles (28 days each, 21 days with tablet intake followed by a 7-day tablet-free interval) one post-treatment cycle
Assessment of cervical mucus according to Insler | 4 cycles: one cycle before treatment followed by two treatment cycles (28 days each, 21 days with tablet intake followed by a 7-day tablet-free interval) one post-treatment cycle
Pharmacokinetic evaluation in volunteers who receive SH T04769G | 4 cycles: one cycle before treatment followed by two treatment cycles (28 days each, 21 days with tablet intake followed by a 7-day tablet-free interval) one post-treatment cycle

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany